CLINICAL TRIAL: NCT04574687
Title: Effects of Action Observation Therapy on Fine Motor Skills of Upper Limb Functions in Chronic Stroke Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/LHR//19/029 Sidra Sikander
Record Dates: First submitted 2020-09-25; First posted 2020-10-05 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Chronic Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurodevelopmental Techniques (Active Comparator): Conventional treatment protocol including active and active-assissted ROM exercises. (b)Proprioceptive neuro-muscular facilitation techniques. (c)Neuromuscular Developmental Techniques.
  Interventions: Other: Neurodevelopmental Techniques
- Action observation Therapy (Experimental): (a) active range of motion (AROM) exercises (10 min), (b) reaching movement or object manipulation (10 min), and (c) UE functional tasks (15 min). + Conventional treatment protocol as in group A
  Interventions: Other: Action observation Therapy

INTERVENTIONS:
Other: Neurodevelopmental Techniques — )Conventional treatment protocol including active and active-assissted ROM exercises. (b)Proprioceptive neuro-muscular facilitation techniques. (c)Neuromuscular Developmental Techniques.
  Arms: Neurodevelopmental Techniques
Other: Action observation Therapy — (a) active range of motion (AROM) exercises (10 min), (b) reaching movement or object manipulation (10 min), and (c) UE functional tasks (15 min). + Conventional treatment protocol as in group A
  Arms: Action observation Therapy

SUMMARY:
This study will be conducted to evaluate the outcomes of action observation therapy on fine motor skills of affected upper limb among patients with chronic stroke.

DETAILED DESCRIPTION:
The data for study will be collected for the duration of 5 months, data will be collected at 1st, 4th, 8th, 12th and then at 16th week of follow up. It is a Randomized Control Trial. Patients will be selected by Consecutive Sampling from Ittefaq Hospital Trust, Lahore. All patients were right handed prior to stroke. Screening tools used will be Canadian Neurological Scale, the Mini-Mental State Examination (MMSE), the Bell Barrage test, and the ideomotor apraxia test (SpinnlerRognoni).Tests for assessment will be Fugl-Meyer test (FM) (of the upper limb), Frenchay Arm test (FAT), Box and Block test (BBT), Modified Ashworth Scale (AS) and Functional Independence Measure Motor items (FIMM). The SPSS version 21 will be used for analyzing data. The descriptive data will be expressed in Frequency and Percentages, while within the group differences will be measured by Mixed Model Anova.

ELIGIBILITY:
Inclusion Criteria:

* First-ever stroke,
* Enrolled 6 months after the event onset with ischemia or primary hemorrhage.
* All patients were right handed prior to stroke.

Exclusion Criteria:

* Posterior circulation infarction,
* Subarachnoid hemorrhage,
* Severe forms of neglect and anosognosia (number of errors in Bell Barrage test≥15)
* Impaired comprehension (Token test score ≤ 17)
* History of endogenous depression or serious psychiatric disorders, and
* Severe visual deficits (restricting the access to visual stimuli).

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-28 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA): | 2 months
  Scoring. The Fugl-Meyer Assessment scale is an ordinal scale that has 3 points for each item. A zero score is given for the item if the subject cannot do the task. A score of 1 is given when the task is performed partially and a score of 2 is given when the task is performed fully.
Box and Block Test (BBT) | 2 months
  Scoring The score is the number of blocks carried from one compartment to the other in one minute. Score each hand separately.
Frenchay Arm Test (FAT): | 2months
  The Frenchay Arm Test (FAT) is devised for measuring the motor control in proximal joints and dexterity of the upper limb during ADL performance in patients with impairments caused by neurological conditions.Scoring and Score Interpretation Each item is scored as either pass (=1) or fail (=0). Total scores range from 0 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Shabbir, Phd, Principal Investigator — Riphah International University
Locations (1):
- Riphah IU, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee D, Roh H, Park J, Lee S, Han S. Drinking behavior training for stroke patients using action observation and practice of upper limb function. J Phys Ther Sci. 2013 May;25(5):611-4. doi: 10.1589/jpts.25.611. Epub 2013 Jun 29. PMID 24259813
- [Background] Sugg K, Muller S, Winstein C, Hathorn D, Dempsey A. Does Action Observation Training With Immediate Physical Practice Improve Hemiparetic Upper-Limb Function in Chronic Stroke? Neurorehabil Neural Repair. 2015 Oct;29(9):807-17. doi: 10.1177/1545968314565512. Epub 2015 Jan 22. PMID 25613984
- [Background] Franceschini M, Agosti M, Cantagallo A, Sale P, Mancuso M, Buccino G. Mirror neurons: action observation treatment as a tool in stroke rehabilitation. Eur J Phys Rehabil Med. 2010 Dec;46(4):517-23. Epub 2010 Apr 23. PMID 20414184
- [Background] Sale P, Franceschini M. Action observation and mirror neuron network: a tool for motor stroke rehabilitation. Eur J Phys Rehabil Med. 2012 Jun;48(2):313-8. Epub 2012 Apr 20. PMID 22522432
- [Background] Franceschini M, Ceravolo MG, Agosti M, Cavallini P, Bonassi S, Dall'Armi V, Massucci M, Schifini F, Sale P. Clinical relevance of action observation in upper-limb stroke rehabilitation: a possible role in recovery of functional dexterity. A randomized clinical trial. Neurorehabil Neural Repair. 2012 Jun;26(5):456-62. doi: 10.1177/1545968311427406. Epub 2012 Jan 10. PMID 22235059
- [Background] Johansson BB. Current trends in stroke rehabilitation. A review with focus on brain plasticity. Acta Neurol Scand. 2011 Mar;123(3):147-59. doi: 10.1111/j.1600-0404.2010.01417.x. Epub 2010 Aug 19. PMID 20726844
- [Background] Garrison KA, Winstein CJ, Aziz-Zadeh L. The mirror neuron system: a neural substrate for methods in stroke rehabilitation. Neurorehabil Neural Repair. 2010 Jun;24(5):404-12. doi: 10.1177/1545968309354536. Epub 2010 Mar 5. PMID 20207851
- [Background] Han C, Wang Q, Meng PP, Qi MZ. Effects of intensity of arm training on hemiplegic upper extremity motor recovery in stroke patients: a randomized controlled trial. Clin Rehabil. 2013 Jan;27(1):75-81. doi: 10.1177/0269215512447223. Epub 2012 Jul 16. PMID 22801472
- [Background] Eng K, Siekierka E, Pyk P, Chevrier E, Hauser Y, Cameirao M, Holper L, Hagni K, Zimmerli L, Duff A, Schuster C, Bassetti C, Verschure P, Kiper D. Interactive visuo-motor therapy system for stroke rehabilitation. Med Biol Eng Comput. 2007 Sep;45(9):901-7. doi: 10.1007/s11517-007-0239-1. Epub 2007 Aug 9. PMID 17687578
- [Background] Ertelt D, Small S, Solodkin A, Dettmers C, McNamara A, Binkofski F, Buccino G. Action observation has a positive impact on rehabilitation of motor deficits after stroke. Neuroimage. 2007;36 Suppl 2:T164-73. doi: 10.1016/j.neuroimage.2007.03.043. Epub 2007 Mar 31. PMID 17499164
- [Derived] Borges LR, Fernandes AB, Oliveira Dos Passos J, Rego IAO, Campos TF. Action observation for upper limb rehabilitation after stroke. Cochrane Database Syst Rev. 2022 Aug 5;8(8):CD011887. doi: 10.1002/14651858.CD011887.pub3. PMID 35930301